## The Effect of Different Exercise Types on Migraine Frequency in Individuals with Migraine

NCT05568004

This is the preplanned and the primary analysis of these data. There were no missing data. Statistical analysis was conducted by a researcher blinded to the participants' groups using the Statistical Package for Social Sciences (SPSS) version 26.0 (IBM Corp., Armonk, NY, USA). The Shapiro–Wilk test and histograms evaluated the data for normal distribution, and the Levene test confirmed homogeneous variances between groups (p > 0.05). Continuous data following a normal distribution are presented as mean  $\pm$  standard deviation (SD). The independent samples t test or Mann–Whitney U test was used to compare independent continuous data between groups, while the chi-square or Fisher's exact test was used to compare categorical data. Friedman two-way ANOVA was used to analyze dependent variables, while the two-way mixed ANOVA was used to examine the changes between groups over time. Before the two-way mixed ANOVA, boxplot evaluation confirmed no outliers. Mauchly's sphericity test showed that the assumption of sphericity for two-way interaction was met. Tukey's correction was used for pairwise subgroup comparisons. A p-value of < 0.05 was considered statistically significant for all analyses.